CLINICAL TRIAL: NCT04086238
Title: An Open-Label, Randomized, Four-Period, Three-Block, Pharmacokinetic Study of Three Formulations of Decitabine/Tetrahydrouridine (THU) Combination Modified Release Capsules in Healthy Adults Under Fasting and Fed Conditions
Brief Title: Effect of Food on the Pharmacokinetics of Decitabine/Tetrahydrouridine Combination Capsules in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpiDestiny, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EPI01-CP.002
Record Dates: First submitted 2019-09-10; First posted 2019-09-11 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2019-09

CONDITIONS: Healthy
MeSH Terms: interventions — Decitabine; Tetrahydrouridine

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, three-block, four-period study to evaluate the relative pharmacokinetics of three test formulations of decitabine and THU in a modified release THU and decitabine combination capsule (EPI01) in healthy male and female adults
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Formulation A Fasted (Other): EPI01 Formulation A (moderate release): 3 capsules each containing decitabine (5 mg) and THU (250 mg) administered under fasting conditions. Single oral administration with 250mL of water.
  Interventions: Drug: Decitabine
- Formulation A Fed (Experimental): EPI01 Formulation A (moderate release): 3 capsules each containing decitabine (5 mg) and THU (250 mg) administered under fed conditions. Single oral administration with 250mL of water.
  Interventions: Drug: Decitabine
- Formulation B Fasted (Other): EPI01 Formulation B (slow reelase): 3 capsules each containing decitabine (5 mg) and THU (250 mg) administered under fasting conditions. Single oral administration with 250mL of water.
  Interventions: Drug: Decitabine
- Formulation B Fed (Experimental): EPI01 Formulation B (slow release): 3 capsules each containing decitabine (5 mg) and THU (250 mg) administered under fed conditions. Single oral administration with 250mL of water.
  Interventions: Drug: Decitabine
- Formulation C Fasted (Other): EPI01 Formulation C (retarded release): 3 capsules each containing decitabine (5 mg) and THU (250 mg) administered under fasting conditions. Single oral administration with 250mL of water.
  Interventions: Drug: Decitabine
- Formulation C Fed (Experimental): EPI01 Formulation C (retarded release): 3 capsules each containing decitabine (5 mg) and THU (250 mg) administered under fed conditions. Single oral administration with 250mL of water.
  Interventions: Drug: Decitabine

INTERVENTIONS:
Drug: Decitabine — Capsules containing a combination of decitabine and THU
  Other Names: EPI01; Tetrahydrouridine

SUMMARY:
This study is to investigate the effect of a high fat meal on the pharmacokinetics of decitabine and THU in healthy adults when administered as a modified release formulation of the 2 drugs in combination.

DETAILED DESCRIPTION:
This study is to evaluate the relative pharmacokinetics of oral decitabine and tetrahydrouridine (THU) after a high-fat, high-calorie (FDA standard) meal as compared to decitabine and THU under fasting conditions in healthy adult male and female subjects. In addition, this study is to compare the pharmacokinetic parameters between male and female subjects, and also to capture safety information for the decitabine and THU combination in healthy subjects after oral dosing.

ELIGIBILITY:
Inclusion Criteria:

* Understands and voluntarily signs a written Informed Consent Form prior to any study related procedures being performed and is able to adhere to restrictions and examination schedules.
* Able to communicate with the investigator, and to understand and comply with the requirements of the study.
* A healthy male or female from any race between 18 to 50 years of age (inclusive). If female, she meets at least one of the following criteria: Surgically sterile (hysterectomy, tubal ligation or bilateral oophorectomy); Or ≥1 year postmenopausal (will have a follicle-stimulating hormone test performed at screening to confirm postmenopausal status)
* A body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and a minimum weight of 50 kg at screening.
* Subjects must be free of any clinically significant disease that would interfere with the study evaluations, and be in good health as determined by past medical history, physical examination, and ECG at screening.
* Vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the supine position after the subject has rested for at least 5 minutes. At screening, the potential subject must be afebrile, with a systolic blood pressure between 90 and 140 mmHg (inclusive), diastolic blood pressure between 60 and 90 mmHg (inclusive), and pulse rate between 50 and 100 bpm (inclusive).
* Male subjects (including those who have had a documented vasectomy) must use a double-barrier local contraception (i.e., spermicidal gel plus condom) when engaging in sexual activity with women of childbearing potential while on study medication and for 28 days after the last dose of study medication. They must also agree to refrain from sperm donations while on study drug, for the entire duration of the study, and for at least 28 days after the last dose of study drug.

Exclusion Criteria:

* History (within 3 years prior to screening) or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, oncologic, or psychiatric disease or any other condition, including the presence of laboratory abnormalities, that, in the opinion of the Investigator, would jeopardize the safety of the subject or the validity of the study results.
* Any serious medical condition, clinically significant laboratory abnormality, or psychiatric illness that would prevent the subject from signing the Informed Consent Form.
* Used any prescribed systemic or topical medication within 30 days of the first dose administration.
* Used any non-prescribed systemic (including herbal medicines, e.g. St. John's Wort) or topical medication within 7 days of the first dose administration (with the exception of vitamin/mineral supplements)
* Subjects who have any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism and excretion (ADME), including a past cholecystectomy.
* Exposed to an investigational drug (new chemical entity) within 90 days preceding the first dose administration or currently enrolled in any investigational trials.
* Donated blood or plasma within 8 weeks preceding the first dose administration.
* History of multiple drug allergies.
* Any clinically significant allergic disease (excluding nonactive hayfever).
* History of drug abuse within 2 years prior to dosing, or a positive drug test at screening or either check-in.
* History of alcohol abuse within 2 years prior to dosing, or a positive alcohol test at screening or either check-in.
* Smokers or users of other tobacco products (e.g., chewing tobacco, or those using nicotine-containing products (i.e., patches, gum) within 3 months prior to screening, or a positive urine cotinine test at screening or either check-in.
* Known to have serum hepatitis or known to be a carrier of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody, or tests positive for HIV (human immunodeficiency virus) antibodies at screening.
* Subject must not consume beverages and foods containing grapefruit, broccoli, poppy seeds, Brussels sprouts, pomegranate, star fruit, char-grilled meat, or caffeine/xanthine from 48 hours prior to the first dose of study medication until the end-of-study visit. Subjects will be instructed not to consume any of the above products; however, allowance for an isolated single incidental consumption may be evaluated and approved by the study investigator based on the potential for interaction with the study drug.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
Absorption of Decitabine | 24 hours
  Area under the concentration-time curve (AUC) from time of dosing to the last quantifiable concentration of Decitabine
Decitabine plasma concentration | 24 hours
  Maximum concentration (Cmax) of Decitabine in plasma
Absorption of Tetrahydrouridine | 24 hours
  Area under the concentration-time curve (AUC) from time of dosing to the last quantifiable concentration of THU

SECONDARY OUTCOMES:
Safety of decitabine and tetrahydrouridine | 24 hours
  The number of subjects reporting adverse events such as nausea and headache.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia A Zamora, MD, Principal Investigator — Worldwide Clinical Trails Early Phase Services, LLC
Locations (1):
- Worldwide Clinical Trial, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Undecided